CLINICAL TRIAL: NCT03107520
Title: Use of Intraoperative Contrast-enhanced Ultrasound to Evaluate Femoral Head Perfusion in Infants With Developmental Dysplasia of the Hip at the Time of Surgical Reduction
Brief Title: Intraoperative Contrast-Enhanced Ultrasound Evaluation of Blood Flow at the Time of Surgical Hip Reduction for DDH
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Bracco Diagnostics, Inc (Industry); Pediatric Orthopaedic Society of North America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-013583
Record Dates: First submitted 2017-03-23; First posted 2017-04-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Developmental Dysplasia of the Hip
Keywords: contrast-enhanced ultrasound; Lumason; developmental dysplasia of the hip (DDH); avascular necrosis
MeSH Terms: conditions — Developmental Dysplasia of the Hip; Osteonecrosis

STUDY DESIGN:
Masking Description: The surgeon and musculoskeletal radiologist administering the contrast-enhanced ultrasound will not be blinded at the time of the intervention; however, they will be blinded when comparing the results of the CEUS to standard-of-care perfusion MRI and 3-years postop radiographs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DDH Surgical Reduction Patients (Experimental): Infants treated for DDH who failed conservative measures and are undergoing intraoperative open or closed hip reduction. Intraoperative contrast-enhanced ultrasound using Lumason contrast agent will be administered to improve visualization of the epiphyseal vascularity after hip reduction and during placement of the spica cast.
  Interventions: Diagnostic Test: Intraoperative contrast-enhanced ultrasound (CEUS); Drug: Lumason

INTERVENTIONS:
Diagnostic Test: Intraoperative contrast-enhanced ultrasound (CEUS) — An intraoperative CEUS of the dysplastic femoral head will be performed after surgical reduction of the femoral head and during placement of the spica cast.
Drug: Lumason — Administration of Lumason contrast agent to improve visualization of epiphyseal vascularity in the femoral head.

SUMMARY:
This study evaluates the feasibility and utility of contrast-enhanced ultrasound to provide real-time assessment of blood flow to the femoral head in infants undergoing surgical reduction for developmental dysplasia of the hip.

DETAILED DESCRIPTION:
For children presenting with late-diagnosed developmental dysplasia of the hip, a closed or open hip reduction followed by hip spica casting may be indicated if conservative treatment fails. Although closed or open reduction and casting is largely successful for relocating a hip, iatrogenic avascular necrosis remains a major source of morbidity as a result of the surgical procedure.

Although recent evidence has demonstrated that postoperative gadolinium-enhanced magnetic resonance (MR) studies may be useful in assessing perfusion of the hip after surgery, these studies are not performed until after the cast is placed and they do not elucidate the specific intraoperative steps that increase risk for osteonecrosis. Contrast-enhanced ultrasound (CEUS) may be a reliable and effective alternative.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 4 months and up to and including 24 months of age at the time of surgery.
* Diagnosed with DDH.
* Failed conservative treatment, or present with late-diagnosed DDH (where conservative treatment would not be appropriate to initiate at their age), and are undergoing closed or open reduction and spica casting.
* Informed consent (parental permission)

Exclusion Criteria:

* > 24 months of age at the time of surgery.
* Subjects with DDH who are successfully treated with conservative measures and do not require surgical reduction.
* Previous open hip reduction of the affected side
* Children with known complex congenital heart disease or unstable cardiopulmonary conditions (as noted in the package labeling for Lumason) including acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure or serious ventricular arrhythmias will be excluded.
* History of allergic reaction to Lumason, sulfur hexafluoride, sulfur hexafluoride lipid microsphere components, or other ingredients in Lumason (polyethylene glycol, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Ns), palmitic acid).Parental/guardian permission (informed consent) and if appropriate, child assent.

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Visualization of epiphyseal vascularity in the femoral head | 1 day
  The visualization of epiphyseal vascularity on the sonogram from intraoperative CEUS will be assessed by a trained sonographer and musculoskeletal radiologist administering the CEUS and reviewing the images.

SECONDARY OUTCOMES:
Comparison of CEUS and Post-Operative Imaging | Approximately 3 years
  The images obtained via intraoperative CEUS will be compared to standard-of-care postoperative perfusion MR imaging and 1-year follow-up radiographs.
Estimate and predict the likelihood of developing avascular necrosis | Approximately 3 years
  To estimate the relationship and predict the likelihood of developing avascular necrosis (outcome variable) and CEUS performance (explanatory variable) as measured by CEUS score

CONTACTS AND LOCATIONS:
Overall Officials: Wudbhav N Sankar, MD, Principal Investigator — Children's Hospital of Philadelphia; Susan Back, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darge K, Papadopoulou F, Ntoulia A, Bulas DI, Coley BD, Fordham LA, Paltiel HJ, McCarville B, Volberg FM, Cosgrove DO, Goldberg BB, Wilson SR, Feinstein SB. Safety of contrast-enhanced ultrasound in children for non-cardiac applications: a review by the Society for Pediatric Radiology (SPR) and the International Contrast Ultrasound Society (ICUS). Pediatr Radiol. 2013 Sep;43(9):1063-73. doi: 10.1007/s00247-013-2746-6. Epub 2013 Jul 11. PMID 23843130
- [Background] Rosenbaum DG, Servaes S, Bogner EA, Jaramillo D, Mintz DN. MR Imaging in Postreduction Assessment of Developmental Dysplasia of the Hip: Goals and Obstacles. Radiographics. 2016 May-Jun;36(3):840-54. doi: 10.1148/rg.2016150159. Epub 2016 Apr 1. PMID 27035836
- [Background] Tiderius C, Jaramillo D, Connolly S, Griffey M, Rodriguez DP, Kasser JR, Millis MB, Zurakowski D, Kim YJ. Post-closed reduction perfusion magnetic resonance imaging as a predictor of avascular necrosis in developmental hip dysplasia: a preliminary report. J Pediatr Orthop. 2009 Jan-Feb;29(1):14-20. doi: 10.1097/BPO.0b013e3181926c40. PMID 19098638
- [Background] Gornitzky AL, Georgiadis AG, Seeley MA, Horn BD, Sankar WN. Does Perfusion MRI After Closed Reduction of Developmental Dysplasia of the Hip Reduce the Incidence of Avascular Necrosis? Clin Orthop Relat Res. 2016 May;474(5):1153-65. doi: 10.1007/s11999-015-4387-6. PMID 26092677